CLINICAL TRIAL: NCT06751355
Title: Precision Imaging to Evaluate Kaposi Sarcoma (PRIME-KS): A Device Feasibility Trial
Acronym: PRIME-KS
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pensievision (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202501193; U01CA292765 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Kaposi Sarcoma
Keywords: Kaposi; Imaging; Photography; 3D
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SkinScan3D: Consenting and eligible patients will have tumor assessments performed at a single visit. These assessments will be done by ruler or calipers, cell phone 2D photographs, and SS3D camera.
  Interventions: Device: SkinScan3D camera

INTERVENTIONS:
Device: SkinScan3D camera — The SkinScan3D (SS3D) is a portable, battery-powered imaging prototype which can successfully achieve all-focus, 3D images using low-cost, off-the-shelf components.
  Other Names: SS3D

SUMMARY:
While tremendous progress has been made against HIV, both in preventing the infection and in treating AIDS, the disease it causes, AIDS-related malignancies like Kaposi sarcoma (KS) remain a significant health burden, in both the U.S. and especially the developing world. In many cases, multiple KS lesions develop simultaneously, and may progress and regress independently. Photographs are an essential part of the evaluation for KS, as reflected in their formal usage described in the KS Tumor Assessment Manual of Procedures. However, acquiring a clear, informative photo is not trivial, since anatomy is 3D and conventional imaging is 2D. The importance of accurate, quantitative 3D information is especially pronounced for the treatment of KS because when a tumor responds positively to treatment, the initial change is usually a flattening of the lesion, without any significant change in the projected 2D area. To evaluate the vertical space, along with other characteristics of a KS lesion, we have created an innovative imaging system, SkinScan3D, utilizing new commercial liquid lens technologies and AI based image analysis software, with strategies borrowed from astronomical imaging techniques previously used on NASA space telescopes. In this study, the investigators will develop and demonstrate a protocol for recording measurable 3D parameters, which may be used in a longitudinal study to rigorously monitor therapeutic responses of KS and statistically compare with that of the conventional AMC criteria.

ELIGIBILITY:
Eligibility Criteria:

* Have been diagnosed with histologically or cytologically proven Kaposi sarcoma (KS).
* Has at least 3 cutaneous Kaposi sarcoma lesions.
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will enroll at Siteman Cancer Center at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of capturing 3D images of cutaneous KS lesions | Day 1
  Feasibility is defined as > 90% of lesions captured in the conventional imaging procedures are also seen in the SkinScan3D data and > 70% of lesions detected with SkinScan3D result in a measurable 3D shape not available in the conventional measurement (and quantitative color measurements are achieved for > 90% of such lesions).

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu